CLINICAL TRIAL: NCT04948970
Title: Development of New Technology for One-step Diagnosis of Adrenal Diseases Based on Adrenal Hormone Panel
Brief Title: Steroid Panel for One-step Diagnosis of Adrenal Diseases
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2105-008-1215
Record Dates: First submitted 2021-06-14; First posted 2021-07-02 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2021-06

CONDITIONS: Adrenal Disease
MeSH Terms: conditions — Adrenal Gland Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum, Urine, Saliva, Hair
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to develop a one-step diagnostic method for adrenal diseases, Patients with adrenal diseases including non-functioning adrenal adenoma, adrenal Cushing's syndrome, primary aldosteronism, and pheochromocytoma will be recruited. Using mass spectrometry analysis based on a multisteroid panel, serum, urine, saliva, and hair samples of the patients will be analyzed. The diagnostic yield of each and combination of steroids will be evaluated.

DETAILED DESCRIPTION:
Adrenal diseases consist of heterogenous diseases. To differentiate various adrenal diseases, multiple steps of diagnostic tests are needed. In this study, the investigators aimed to develop a one-step diagnostic method to differentiate various adrenal diseases using multisteroid panel.

About 400 patients with adrenal diseases including non-functioning adenoma, adrenal Cushing's syndrome, primary aldosteronism, and pheochromocytoma will be recruited. Serum, hair, saliva, and urine samples of the patients will be analyzed using mass spectrometry. Each and combination of multisteroid will be evaluated for diagnosing adrenal diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with adrenal diseases

Exclusion Criteria:

* Taking medications that can affect steroid metabolism
* Major depression, chronic alcoholism
* Suspected cancer metastasis to adrenal glands
* Other acute stress conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study subjects will consist of patients who were treated for adrenal diseases such as adrenal incidentaloma, adrenal Cushing's syndrome, primary aldosteronism, and pheochromocytoma at Seoul National University Hospital, and who agreed to participate in this study at Seoul National University Hospital and Seoul National University Bundang Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2021-06-21 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of multisteroid panel for differentiating adrenal diseases | Within 1 year after subject recruitment when the final diagnosis of adrenal diseases are made
  * Evaluate how accurately the developed multisteroid panel diagnoses adrenal disease by measuring sensitivity (%) and specificity (%) for diagnosis of Cushing's syndrome.
  * Evaluate how accurately the developed multisteroid panel diagnoses adrenal disease by measuring sensitivity (%) and specificity (%) for diagnosis of primary aldosteronism.
  * Evaluate how accurately the developed multisteroid panel diagnoses adrenal disease by measuring sensitivity (%) and specificity (%) for diagnosis of pheochromocytoma.

SECONDARY OUTCOMES:
Diagnostic accuracy of each steroid component for differentiating adrenal diseases | Within 1 year after subject recruitment when the final diagnosis of adrenal diseases are made
  Evaluate how accurately each component of the steroid panel differentiate adrenal diseases.
  * Sensitivity (%) and specificity (%) of each steroid measures for adrenal Cushing's syndrome will be calculated.
  * Sensitivity (%) and specificity (%) of each steroid measures for primary aldosteronism will be calculated.
  * Sensitivity (%) and specificity (%) of each steroid measures for pheochromocytoma will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Jung Hee Kim, M.D., Ph.D., Study Chair — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea

IPD SHARING:
Plan to Share IPD: No